CLINICAL TRIAL: NCT00245336
Title: A Phase 3, Randomized, Double-Blind, Controlled, Comparative Efficacy and Safety Study of Topical Recombinant Human Thrombin (rhThrombin) and Thrombin-JMI (Bovine Thrombin) in Surgical Hemostasis
Brief Title: Study of Recombinant Human Thrombin for Bleeding During Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZymoGenetics (Industry)
Responsible Party: Allan Alexander, MD, ZymoGenetics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 499E01
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2009-03-09 (Estimated); Status verified 2009-03

CONDITIONS: Surgical Hemostasis
Keywords: hemostasis; surgery; hemostatics; randomized controlled trial; phase 3
MeSH Terms: interventions — recombinant human thrombin; Thrombin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): rThrombin
  Interventions: Biological: rThrombin
- 2 (Active Comparator): bThrombin
  Interventions: Drug: bovine thrombin

INTERVENTIONS:
Biological: rThrombin — 1000 U/mL applied topically in combination with absorbable gelatin sponge
  Arms: 1
Drug: bovine thrombin — 1000 U/mL applied topically in combination with absorbable gelatin sponge
  Other Names: Thrombin-JMI
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether recombinant human Thrombin (rhThrombin) is effective in stopping bleeding during surgery, in comparison with bovine thrombin.

DETAILED DESCRIPTION:
This is a Phase 3 multiple site, randomized, double-blind, controlled trial designed to evaluate the comparative efficacy and safety of rhThrombin and bovine thrombin in patients undergoing spinal surgery, hepatic resection, peripheral arterial bypass surgery, or arteriovenous graft formation for hemodialysis access.

After establishing eligibility, subjects will be randomized in a 1:1 ratio to receive rhThrombin (1000 U/mL) or bovine thrombin (1000 U/mL). During a surgical procedure, study participants will be treated with blinded study drug (rhThrombin or bovine thrombin) in combination with an absorbable gelatin sponge at appropriate bleeding evaluation site(s) and time to hemostasis (TTH) will be assessed for up to 10 minutes. Bleeding appropriate for TTH evaluation is defined as mild to moderate bleeding, either on its own or remaining after brisk bleeding has been controlled by standard surgical modalities. Blinded study drug may also be used at additional appropriate bleeding sites. Study participants will have follow-up visits at about 2 days and 1 month after surgery. Approximately 400 to 600 patients will participate in the study. The final sample size will be determined based on blinded interim results.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing spinal surgery, hepatic resection, peripheral arterial bypass surgery, or arteriovenous graft formation for hemodialysis access

Exclusion Criteria:

* Subject has undergone a therapeutic surgical procedure within 30 days prior to surgery
* Subject has history of heparin-induced thrombocytopenia
* Subject has known antibodies or hypersensitivity to thrombin or other coagulation factors or known sensitivity to other components of the study treatment
* Subject has received blood products within 24 hours prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Time to hemostasis, as measured by the incidence of hemostasis within 10 minutes | 10 minutes

SECONDARY OUTCOMES:
Incidence and severity of adverse events | Up to 29 days
Incidence and grade of clinical laboratory abnormalities | Up to 29 days
Incidence of anti-product antibodies | Up to 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Reynolds, MD, PhD, Study Director — ZymoGenetics; William Chapman, MD, Principal Investigator — Washington University School of Medicine; Kenneth Renkens, MD, Principal Investigator — Indiana Spine Group; Fred Weaver, MD, Principal Investigator — University of Southern California
Locations (28):
- United States (28):
  - Cardio Thoracic Surgeons, P.C., Birmingham, Alabama
  - Cardio Thoracic Surgeons, P.C., Medical Center East / Baptist Montclair, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Methodist Hospital, Arcadia, California
  - Glendale Adventist Medical Center, Glendale, California
  - University of Southern California, Keck School of Medicine, Los Angeles, California
  - Huntington Memorial Hospital, Pasadena, California
  - Baptist Clinical Research, Pensacola, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Northwestern University Vascular Surgery, Chicago, Illinois
  - Indiana Spine Group, Indianapolis, Indiana
  - Bluegrass Orthopedics/Bluegrass Musculoskeletal Research, Lexington, Kentucky
  - Vascular Surgery Associates, Baton Rouge, Louisiana
  - Tulane University Abdominal Transplant, New Orleans, Louisiana
  - VAMC Clinical Research Center, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Mt. Sinai School of Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of North Texas Science Center at Fort Worth, Fort Worth, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Physician's Research Options, LLC/The Intermountain Spine Institute, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Weaver FA, Lew W, Granke K, Yonehiro L, Delange B, Alexander WA; Study Investigators. A comparison of recombinant thrombin to bovine thrombin as a hemostatic ancillary in patients undergoing peripheral arterial bypass and arteriovenous graft procedures. J Vasc Surg. 2008 Jun;47(6):1266-73. doi: 10.1016/j.jvs.2008.01.034. Epub 2008 Apr 28. PMID 18440754
- [Derived] Chapman WC, Singla N, Genyk Y, McNeil JW, Renkens KL Jr, Reynolds TC, Murphy A, Weaver FA. A phase 3, randomized, double-blind comparative study of the efficacy and safety of topical recombinant human thrombin and bovine thrombin in surgical hemostasis. J Am Coll Surg. 2007 Aug;205(2):256-65. doi: 10.1016/j.jamcollsurg.2007.03.020. Epub 2007 Jun 27. PMID 17660072